CLINICAL TRIAL: NCT06747390
Title: A Phase I Randomized Controlled Trial of Intratumoral Lidocaine Injection Before Transoral Robotic Surgery (TORS) and Neck Dissection for HPV-Associated Oropharyngeal Squamous Cell Carcinoma
Brief Title: Intratumoral Lidocaine Injection Before Oropharyngeal Cancer Surgery
Acronym: 856397
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ryan Carey (Other)
Responsible Party: Sponsor-Investigator, Ryan Carey, Assistant Professor, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPCC12324
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma (OPSCCA); Oropharyngeal Cancer; Human Papilloma Virus; Squamous Cell Carcinoma
Keywords: TransOral Robotic Surgery (TORS); Oropharyngeal Squamous Cell Carcinoma; Oropharyngeal Cancer; Human Papilloma Virus; Squamous Cell Carcinoma; Lidocaine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Carcinoma, Squamous Cell | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized and blinded to intratumoral injection of 1% lidocaine (intervention arm) or no injection (control arm) at the time of direct laryngoscopy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm - No Injection (No Intervention): No injection at the time of direct laryngoscopy.
- Lidocaine Injectible product (Experimental): Intratumoral injection of 1% lidocaine at the time of direct laryngoscopy.
  Interventions: Drug: Lidocaine 1% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — 1% lidocaine will be injected under direct visualization (not exceeding the maximum tolerated dose of 4.5 mg/kg body weight) into the primary tumor with the aim to distribute the lidocaine evenly into the tumor.
  Arms: Lidocaine Injectible product

SUMMARY:
Based on evidence that the local anesthetic lidocaine may have anticancer effects, this study will assess the safety and efficacy of intratumoral lidocaine injection at the time of direct laryngoscopy prior to TransOral Robotic Surgery (TORS) and neck dissection for oropharyngeal squamous cell carcinoma (OPSCC). The primary objective of the study is to determine if intratumoral lidocaine injection is safe and causes a major pathologic treatment effect in the primary tumor following surgical resection. The secondary objectives will be to determine if intratumoral lidocaine injection improves locoregional control rates, progression-free survival, metastasis-free survival, and overall survival compared to no injection.

DETAILED DESCRIPTION:
This is a phase I patient-blinded, randomized controlled trial evaluating intratumoral lidocaine injection prior to definitive surgery in HPV associated OPSCC. Patients with OPSCC undergoing direct laryngoscopy who are being considered for definitive TORS and selective neck dissection, will be eligible. Patients will be randomized and blinded to intratumoral injection of 1% lidocaine (intervention arm) or no injection (control arm) at the time of direct laryngoscopy. After administration of general anesthesia and biopsy, lidocaine will be injected under direct visualization (not exceeding the maximum tolerated dose of 4.5 mg/kg body weight) into the primary tumor.

Blood samples will be obtained prior to direct laryngoscopy/study intervention (pre-biopsy) and again after the intervention (post-biopsy). Following direct laryngoscopy/study intervention, patients will receive institutional standard of care treatment which may include primary surgery (TORS primary site resection, selective neck dissection, and any indicated adjuvant therapy) or primary radiation (with or without chemotherapy). For patients undergoing surgery, the pathological tumor response (pTR) rate (defined as the area with pathologic response/area pathologic response plus viable tumor) will be determined by the designated study pathologist using increments of 10% for the biopsy and surgery specimens. The scores will be grouped as pTR-0 (<10%), pTR-1 (10%-49%), and pTR-2 (≥50%).

All enrolled patients will be assessed for safety measured by adverse events. If a patient does not ultimately receive primary surgery following their direct laryngoscopy/study intervention (based on surgical candidacy, patient preference, or other reasons), then they will not be counted as an evaluable subject, as the primary endpoint pTR requires a surgical specimen for evaluation. If a patient is determined to have a pathology other than HPV associated OPSCC after their direct laryngoscopy, then they will not be counted as an evaluable subject. The enrollment target will be 30 evaluable subjects.

Primary Objectives: Determine if intratumoral 1% lidocaine injection at the time of direct laryngoscopy prior to TORS and neck dissection for HPV associated OPSCC is safe and causes a major pathologic treatment effect.

Secondary Objectives: Determine if intratumoral 1% lidocaine injection at the time of direct laryngoscopy prior to TORS and neck dissection for HPV associated OPSCC improves the locoregional control rates, progression-free survival, metastasis-free survival, and overall survival compared to no injection.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years older or more.

Histologically confirmed diagnosis of squamous cell carcinoma of the oropharynx or neck.

Clinical T1, T2, T3, or T4 stage disease of the oropharynx (per AJCC 8th Ed).

Any clinical N stage disease (per AJCC 8th Ed).

Patients must be undergoing direct laryngoscopy +/- biopsy at the University of Pennsylvania as part of their work-up for consideration of definitive TORS and selective neck dissection.

Patients must sign an informed consent document that indicates they are aware of the investigational nature of the treatment in this protocol as well as the potential risks and benefits.

Ability to understand and the willingness to provide written informed consent.

---

Exclusion Criteria:

Prior external beam radiation therapy to the head and neck.

Prior chemotherapy for head and neck cancer.

Tumor invades lateral pterygoid muscle, pterygoid plates, lateral nasopharynx, or skull base or encases carotid artery (i.e. AJCC 7th Ed. T4b for OPSCC).

Presence of distant metastatic disease.

Uncontrolled inter-current illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, connective tissue disease or psychiatric illness/social situations that would limit compliance with study requirements.

Known history of hypersensitivity to lidocaine or other amide local anesthetics.

Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of adverse events. | 2 years
  Adverse events (AE) and Serious Adverse Events (SAE) will use the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The CTCAE v.5 utilizes a five point scale to report AEs, defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Pathological tumor response (pTR) in the primary tumor following surgical resection. | 2 years
  The pathological tumor response (pTR) rate (defined as the area with pathologic response/area pathologic response plus viable tumor) will be determined by the designated study pathologist using increments of 10% for the biopsy and surgery specimens. The scores will be grouped as pTR-0 (<10%), pTR-1 (10%-49%), and pTR-2 (≥50%).

SECONDARY OUTCOMES:
2-year locoregional control rates. | 2 years
  Locoregional control is defined as control at the primary site and in the neck.
2-year progression-free survival. | 2 years
  Progression-free survival is defined as the length of time during and after treatment that a patient lives with the disease but it does not get worse.
2-year metastasis-free survival. | 2 years
  Metastasis-free survival is the length of time from the start of treatment for a disease until the patient remains alive without the development of distant metastatic disease.
2-year overall survival. | 2 years
  Overall survival is defined as the length of time from the start of treatment for a disease that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Carey, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller ZA, Mueller A, Kim T, Jolivert JF, Ma RZ, Muthuswami S, Park A, McMahon DB, Nead KT, Carey RM, Lee RJ. Lidocaine induces apoptosis in head and neck squamous cell carcinoma through activation of bitter taste receptor T2R14. Cell Rep. 2023 Dec 26;42(12):113437. doi: 10.1016/j.celrep.2023.113437. Epub 2023 Nov 22. PMID 37995679
- [Background] Carey RM, McMahon DB, Miller ZA, Kim T, Rajasekaran K, Gopallawa I, Newman JG, Basu D, Nead KT, White EA, Lee RJ. T2R bitter taste receptors regulate apoptosis and may be associated with survival in head and neck squamous cell carcinoma. Mol Oncol. 2022 Apr;16(7):1474-1492. doi: 10.1002/1878-0261.13131. Epub 2021 Dec 14. PMID 34717036
- [Background] Badwe RA, Parmar V, Nair N, Joshi S, Hawaldar R, Pawar S, Kadayaprath G, Borthakur BB, Rao Thammineedi S, Pandya S, Balasubramanian S, Chitale PV, Neve R, Harris C, Srivastava A, Siddique S, Vanmali VJ, Dewade A, Gaikwad V, Gupta S. Effect of Peritumoral Infiltration of Local Anesthetic Before Surgery on Survival in Early Breast Cancer. J Clin Oncol. 2023 Jun 20;41(18):3318-3328. doi: 10.1200/JCO.22.01966. Epub 2023 Apr 6. PMID 37023374

DOCUMENTS (1):
  • Study Protocol (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT06747390/Prot_001.pdf